CLINICAL TRIAL: NCT00020878
Title: Celecoxib for Chemoprevention of Primary Lung Cancer
Brief Title: Celecoxib in Preventing Non-Small Cell Lung Cancer in Tobacco Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000068727; UCLA-0012067; NCI-G01-1966
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2016-03

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study (Experimental): See intervention description.
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib — Dosing will occur for a total of 6 months. 400 mg by mouth twice daily.
  Other Names: Celebrex

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. Celecoxib may be effective in preventing lung cancer in tobacco smokers.

PURPOSE: Phase II trial to study the effectiveness of celecoxib in preventing non-small cell lung cancer in tobacco smokers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and feasibility of celecoxib for chemoprevention of primary non-small cell lung cancer in high-risk tobacco smokers.
* Determine the safety and long-term side effects of this drug in this population.

OUTLINE: Patients receive oral celecoxib twice daily for 6 months.

Patients are followed at 2 weeks and then at 6 months.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 45
* Smoked > 20 pack years

Exclusion Criteria:

* Concurrent use of NSAIDs
* Hypersensitivity to celecoxib
* Documented allergic-type reaction to sulfonamides
* History of allergic reaction, urticaria or asthma to aspirin or other NSAIDs
* History of liver dysfunction
* Hypertension or cardiac conditions aggravated by fluid retention and edema
* Previous history of gastrointestinal ulceration, bleeding, or perforation
* Renal dysfunction
* End stage respiratory disease
* Unstable angina
* Other malignancy
* Pregnancy
* Concurrent use of medication known to alter or be affected by alteration of the hepatic p450 2C9 and 2D6 enzymes
* Patents with concurrent medical conditions that may interfere with completion of tests, therapy, or the follow up schedule

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2001-03; Primary Completion 2002-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the expression of Cox-2 and PGE2 in the lungs of tobacco smokers. | 1 year
Evaluate the capacity for an oral Cox-2 inhibitor (Celecoxib) to suppress the intrapulmonary formation of PGE2 | 1 year

SECONDARY OUTCOMES:
Determine the effects of Cox-2 inhibition on biomarkers of field cancerization on histopathologic abnormalities in patients at risk for primary NSCLC | 2 years
Study the potential role of PGE2 and its regulation by Cox-2 specific inhibitors on antitumor immunity within the lung microenvironment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jenny T. Mao, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States